CLINICAL TRIAL: NCT04903054
Title: Selective CD28 Blockade With Lulizumab Compared to CNI Inhibition With Tacrolimus in Renal Transplant Recipients
Brief Title: Selective CD28 Blockade in Renal Transplant Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited period of availability of a supply of the study drug and difficulties in enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT RTB-011; U01AI138909 (NIH); NIAID CRMS ID#: 38687 (Other: DAIT NIAID)
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Kidney Transplantation; Renal Transplant Recipients
Keywords: CD28 blockade; Cluster of Differentiation (CD); CNI inhibition; immune modulation; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — lulizumab pegol; Tacrolimus; thymoglobulin; Antilymphocyte Serum; Methylprednisolone; Adrenal Cortex Hormones; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lulizumab + SOC (Experimental): N=27 participants will receive a loading dose of lulizumab on Day 0, the day of surgery. This will be followed by a maintenance dose administered on a weekly basis (weeks 1 through 26 post-transplant), followed by administration every two weeks (weeks 28 through 52 post-transplant). Method of administration: subcutaneously. Dose unit of measure: milligrams (mgs).
  Plus (+) Standard of Care (SOC) Regimen, per protocol-
  Renal transplant recipients will receive FDA-approved, immunosuppressive medications according to standard of care at Emory Transplant Center:
  * Induction Thymoglobulin: Administered intravenously, dose unit of measure: mgs.
  * Induction Methylprednisolone: Administered intravenously, dose unit of measure: mgs.
  * Maintenance: Mycophenolate mofetil (MMF) administered by mouth twice daily, dose unit of measure: mgs.
  * Maintenance: Beginning the day after methylprednisolone is completed, prednisone will be administered by mouth daily, dose unit of measure: mgs.
  Interventions: Biological: Lulizumab; Biological: Thymoglobulin®; Drug: Methylprednisolone; Drug: Mycophenolate Mofetil; Drug: Prednisone
- Tacrolimus + SOC (Active Comparator): N=27 participants will receive tacrolimus initiated according to local standard of care and adjusted over time (maintenance) to target optimal trough levels measured in ng/mL: 0 to 6 months, 7 to 12 months and, thereafter, until completion of study participation. Dose unit of measure: mg/kg.
  Plus (+) Standard of Care (SOC) Regimen, per protocol-
  Renal transplant recipients will receive FDA-approved, immunosuppressive medications according to standard of care at Emory Transplant Center:
  * Induction Thymoglobulin: Administered intravenously, dose unit of measure: mgs.
  * Induction Methylprednisolone: Administered intravenously, dose unit of measure: mgs.
  * Maintenance: Mycophenolate mofetil (MMF) administered by mouth twice daily, dose unit of measure: mgs.
  * Maintenance: Beginning the day after methylprednisolone is completed, prednisone will be administered by mouth daily, dose unit of measure: mgs.
  Interventions: Drug: Tacrolimus; Biological: Thymoglobulin®; Drug: Methylprednisolone; Drug: Mycophenolate Mofetil; Drug: Prednisone

INTERVENTIONS:
Biological: Lulizumab — Lulizumab is a pegylated, humanized monovalent domain antibody construct that is specific for human cluster of differentiation CD28.
  Other Names: BMS-931699; anti-CD28 domain antibody (anti-CD28 dAb)
  Arms: Lulizumab + SOC
Drug: Tacrolimus — Standard of Care: Renal transplant rejection prophylaxis.
  Other Names: Prograf®
  Arms: Tacrolimus + SOC
Biological: Thymoglobulin® — Standard of Care: Renal transplant rejection prophylaxis.
  Other Names: antithymocyte globulin
Drug: Methylprednisolone — Standard of Care: Renal transplant rejection prophylaxis.
  Other Names: corticosteroid
Drug: Mycophenolate Mofetil — Standard of Care: Renal transplant rejection prophylaxis.
  Other Names: MMF; CellCept®
Drug: Prednisone — Standard of Care: Renal transplant rejection prophylaxis.
  Other Names: corticosteroid

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of lulizumab, a CD28-specific domain antibody (CD28 dAb), compared to tacrolimus, as the primary immunosuppressant in first-time renal transplant recipients.

DETAILED DESCRIPTION:
This is a phase 2a, open-label, prospective, randomized (1:1), controlled, single center study evaluating the safety and efficacy of lulizumab (a CD28 specific domain antibody [CD28dAb]) compared to tacrolimus as the primary immunosuppressant in first-time renal transplant recipients. The study will take place at Emory University Hospital in Atlanta, Georgia, United States (US).

There are two arms/groups in this study, the Control (tacrolimus) group and the Investigational (lulizumab) group. The two arms will be assigned to treatment regimens for the first 12 months after transplantation; at that point, all participants in each arm will be transitioned to a physician directed Standard of Care (SOC) immunosuppressive regimen, and all participants will be assessed at 15 months after transplantation.

All participants will receive induction therapy with Thymoglobulin and Methylprednisolone and maintenance therapy with Mycophenolate Mofetil (MMF) and Prednisone.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Must be able to understand and provide informed consent;
2. Negative crossmatch (actual or virtual) or a Panel Reactive Antibody (PRA) of 0% on historic and admission sera;
3. First time renal transplant from either a living or deceased donor;
4. Deceased donor recipients only: Deceased donor kidneys with Kidney Donor Profile Indices (KDPI) <85%;
5. Female study participants of childbearing potential must have a negative pregnancy test prior to randomization;
6. Agreement to use contraception; according to the Food and Drug Administration (FDA) Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80 percent effective.

   --Female study participants of child-bearing potential and male study participants must consult with their physician and determine the most suitable method(s) from this list to be used from the time that study treatment begins until after study completion;
7. Study participants must have a negative purified protein derivative (PPD) or negative testing for tuberculosis using an approved interferon-gamma release assay (IGRA) blood test, such as:

   * QuantiFERON®-TB Gold In-Tube test (QFT-GIT) or
   * TSPOT® TB test ---PPD or IGRA testing must be documented to have been performed within 52 weeks before transplant;
8. Documented completion of varicella vaccination series ≥ 8 weeks prior to enrollment, OR verification of a history of varicella or zoster by a physician OR positive laboratory confirmation of varicella immunity or disease; and,
9. Immunizations are up-to-date based on the CDC° adult vaccination recommendations:

https://www.cdc.gov/vaccines/schedules/hcp/imz/adult.html

--°Centers for Disease Control and Prevention (CDC)

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness of a study participant to give written informed consent or comply with study protocol;
2. Recipient of previous organ transplant of any type;
3. Need for multi-organ transplant;
4. Calculated panel reactive antibody (cPRA) or panel reactive antibody (PRA) >20% at any time prior to enrollment;
5. Known hypersensitivity to mycophenolate mofetil (MMF) or any of the drug's components;
6. Human immunodeficiency virus (HIV): individuals known to be HIV positive;
7. Known history of Bacillus Calmette-Guérin (BCG) vaccination;
8. Individuals at significant risk of early recurrence of the primary renal disease including: -Focal Segmental Glomerulosclerosis (FSGS)

   * Membranoproliferative Glomerulonephropathy (MPGN) type 2
   * Hemolytic Uremia Syndrome/Thrombotic thrombocytopenic purpura (HUS/TTP), or
   * any other disease that, in the opinion of the investigator, is at increased likelihood of recurrence and which may result in rapid decline in renal function
9. Known history of high-risk thrombotic events or risk factors; including any of the following:

   * Factor V Leiden, elevated homocysteine, positive lupus anticoagulant, elevated anticardiolipin antibody, heparin induced thrombocytopenia
   * A family history of a heritable thrombotic condition
   * Recurrent Deep vein thrombosis (DVT) or Pulmonary Embolism (PE), or
   * Unexplained stillborn infant or recurrent spontaneous abortion of other congenital or acquired thrombotic disorder
10. History of malignancy within 5 years of enrollment or any history of hematogenous malignancy or lymphoma.

    --Note: Study participants with curatively treated non-melanomatous skin cancer or curatively treated cervical carcinoma in situ may be enrolled;
11. Study participants who are on biologic treatments for autoimmune disease;
12. Study participants who are involuntarily detained (e.g. prison, jail, compulsory psychiatric or medical therapy);
13. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator:

    * May pose additional risks from participation in the study,
    * May interfere with the study participant's ability to comply with study requirements, or
    * May impact the quality or interpretation of the data obtained from the study;
14. Human leukocyte antigen (HLA) identical donor/recipient pairing;
15. Use of investigational drugs within 4 weeks of transplant;
16. Study participants who are NOT Epstein-Barr virus (EBV) seropositive

    -A prior documented EBV seropositive result at enrollment does not need to be repeated --For this study, EBV seropositive patients are defined as having evidence of acquired immunity shown by the presence of immunoglobulin G (IgG) antibodies to viral capsid antigen (VCA) and the presence of antibodies to EBV nuclear antigen (EBNA or EBNA1);
17. Hepatitis C virus (HCV): Study participants who are HCV RNA PCR positive at prerandomization re-evaluation

    -Study participants who are seropositive must have 2 consecutive negative HCV RNA PCR at least 24 weeks apart;
18. Hepatitis B virus: Individuals with any of the following are NOT eligible:

    * Recipient or donor positive for hepatitis B surface antigen (HBsAg)
    * Recipient or donor with antibodies to hepatitis B core antigen (anti-HBc)
    * Recipient or donor with HBV DNA detectable by PCR;
19. Recipient of a live or live-attenuated vaccine within 8 weeks prior to transplant;
20. Cytomegalovirus (CMV) seronegative individuals accepting an organ from a CMV seropositive donor;
21. Study participants undergoing transplant using:

    * Organs from donation after circulatory death (DCD) donor
    * Donor with Kidney Donor Profile Index (KDPI) >85%, or
    * Anticipated cold ischemia time >28 hours; or,
22. ABO incompatible donor kidney.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Mean Estimated Glomerular Filtration rate (eGFR) (MDRD) | From Month 2 to Month 12 Post Transplantation
  Efficacy measure. Glomerular Filtration Rate (GFR) will be estimated using the Modification of Diet in Renal Disease (MDRD) equation. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender.

SECONDARY OUTCOMES:
Proportion of Participants Who Remain Free of Biopsy Proven Acute T-Cell Mediated Rejection (aTCMR) | Up to 15 Months Post Transplantation
  Safety measure. Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Proportion of Participants Who Remain Free of Antibody-Mediated Rejection (ABMR) | Up to 15 Months Post Transplantation
  Safety measure. Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Cumulative Incidence of Serious Adverse Events | Up to 15 Months Post Transplantation
  Safety measure.
Incidence of Serious Infection(s) of Special Interest | Up to 15 Months Post Transplantation
  Safety measure. Definition: The occurrence of infection(s) requiring participant hospitalization or prolonged therapy, including but not limited to treatment ≥20 days.
Incidence of Cytomegalovirus (CMV) Viremia | Up to 15 Months Post Transplantation
  Safety measure.
Incidence of BK Polyoma Virus (BKV) Viremia | Up to 15 Months Post Transplantation
  Safety measure.
Incidence of Any Malignancy, Including but Not Limited to PTLD | Up to 15 Months Post Transplantation
  Safety measure.
  Definitions:
  * Malignancy: A term for diseases in which abnormal cells divide without control and can invade nearby tissues.
  * Post-transplant Lymphoproliferative Disorder (PTLD) : A rare but well-known complication of solid organ transplants and hematopoietic stem cell transplantation.
Proportion of Participants Experiencing the Composite Outcome of Death or Allograft Failure | Up to 15 Months Post Transplantation
  Efficacy measure.
Proportion of Participants with Biopsy Proven Acute T-cell Mediated Cellular Rejection (BPaTCMR) | Up to 15 Months Post Transplantation
  Efficacy measure.
  Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Proportion of Participants Treated for Kidney Transplant Rejection | Up to 15 Months Post Transplantation
  Efficacy measure. Definition: Participant requiring treatment for rejection with corticosteroids, T-cell depleting therapy, and/or any other treatment for kidney transplant rejection.
Proportion of Participants Treated for Acute Rejection Due to Clinical Suspicion | Up to 15 Months Post Transplantation
  Efficacy measure. Acute rejection due to a clinical suspicion rather than BPaTCMR or BP-aABMR.
  Definitions:
  * BPaTCMR: Biopsy proven acute T-cell mediated cellular rejection
  * BP-aABMR: Biopsy proven active antibody mediated rejection
Proportion of Participants with Biopsy Proven Active Antibody Mediated Rejection (BP-aABMR) | Up to 15 Months Post Transplantation
  Efficacy measure. Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Proportion of Participants with aTCMR Changes in Allograft Biopsies | Up to 15 Months Post Transplantation
  Efficacy measure.
  Definitions:
  * aTCMR:acute T-cell mediated cellular rejection
  * Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Time to Event for aTCMR Changes in Allograft Biopsies | Up to 15 Months Post Transplantation
  Efficacy measure.
  Definitions:
  * aTCMR:acute T-cell mediated cellular rejection
  * Defined by Banff 2017 kidney criteria.
  Reference: Haas, M. et al. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 18(2):293-307.
Proportion of Participant Who Develop De-Novo Donor Specific Antibody | Up to 15 Months Post Transplantation
  Efficacy measure.
Change in Estimated Glomerular Filtration Rate (eGFR) | From Month 2 to Month 15 Post Transplantation
  Efficacy measure. Glomerular Filtration Rate (GFR) will be estimated using the Modification of Diet in Renal Disease (MDRD) equation. MDRD is an equation (calculation) used to estimate GFR in participants with impaired renal function based on serum creatinine, age, race, and gender.
Proportion of Participants with Delayed Graft Function | Within 1 Month Post Transplantation
  Efficacy measure.
Hemoglobin A1C | Month 12 Post Transplantation
  Efficacy measure. Definition: HbA1c: Glycosylated hemoglobin, a measure of the average plasma concentration of blood sugar (glucose) over the previous three months.
Days to Event: TCMR | Up to 15 Months Post Transplantation
  Efficacy measure. TCMR: T-cell mediated rejection.
Days to Event: Antibody mediated rejection (ABMR) | Up to 15 Months Post Transplantation
  Efficacy measure. ABMR: Antibody mediated rejection.
Days to Event: De-Novo Donor Specific Antibody (DSA) Formation | Up to 15 Months Post Transplantation
  Efficacy measure.
Days to Event: Graft Loss | Up to 15 Months Post Transplantation
  Efficacy measure.
Standardized Blood Pressure | Month 12 and Month 15 Post Transplantation
  Efficacy measure.
Fasting Lipid Profile | Month 12 and Month 15 Post Transplantation
  Efficacy measure. Included: Total cholesterol, LDL, HDL, and triglyceride.

CONTACTS AND LOCATIONS:
Overall Officials: Christian P. Larsen, MD, DPhil, Study Chair — Emory Transplant Center, Emory University; Andrew B. Adams, MD, PhD, Principal Investigator — Emory Transplant Center, Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait